CLINICAL TRIAL: NCT00861055
Title: A Clinical and Microbiological Study of Early Onset Neonatal Sepsis in Refugee Infants and Group B Streptococcal Carriage in Expectant Refugee Mothers Living on the Thai-Burmese Border
Brief Title: Neonatal Sepsis and GBS Carriage Study
Acronym: NSS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU0901
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2016-03

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infants: Infants less than 7 days of age with clinical signs of sepsis
- Mothers: Mothers following antenatal care at SMRU antenatal clinic, Maela camp who are 28 - 30 weeks gestation

SUMMARY:
In the proposed study, the investigators plan to establish the burden of early onset (EO) neonatal sepsis in the newborn population born at Maela Refugee Camp over a two year period.

Aims

1. Define the contribution of Group B streptococcus(GBS) to this problem by establishing:

   * The prevalence of maternal GBS carriage
   * The prevalence of culture positive and culture negative EO GBS sepsis
   * The perinatal risk factors for EO GBS cases
2. Through these data assess the potential for intrapartum antibiotic prophylaxis using different strategies for reducing the burden of neonatal sepsis in this setting
3. To define the serotypes and antibiotic susceptibility profile of carried and invasive GBS strains
4. To evaluate the prevalence of serum antibodies to common GBS capsular serotypes in pregnant women in this population, the influence of carriage on serotype (ST)-specific antibody and the ST-specific antibody concentrations in the mothers of cases of confirmed and clinical GBS disease.

DETAILED DESCRIPTION:
Globally 4 million neonates die each year, the most common cause of death is sepsis. Causes of neonatal sepsis in low and middle income countries are reported to differ from those in the developed world. Gram negative organisms are thought to be more common. Despite group B streptococcus (GBS) carriage rates being apparently similar to the developed world, GBS sepsis is rarely reported in developing countries: our hypothesis is that GBS is an under recognized neonatal pathogen in the developing world. There are many possible explanations why GBS infection may be under reported including wider, less discriminating use of antibiotics in the period just before the onset of labour and inadequate microbiological diagnostic services.

The proposed study, to be conducted at Maela Refugee Camp Thailand, has two components, both being prospective descriptive cohort studies which will be run concurrently:

1. Contribution of GBS to early onset neonatal sepsis at Maela refugee camp
2. GBS carriage, seroepidemiology and GBS antibody study. Infants with neonatal sepsis will be identified clinically. They will be assessed and, after informed consent is taken from their mother, they will have a full septic screen including a complete blood count, serum C-reactive protein, blood culture, lumbar puncture and a deep swab taken from their ear canal. If the ear swab is positive for GBS, and the blood culture is negative for other pathogens, a presumptive diagnosis of EO GBS sepsis will be made. The mother will have 5ml blood sample for GBS serotype-specific antibody testing and a vaginal rectal swab obtained (if this has not been performed already).

Women who consent to take part in the GBS carriage study will, during labour, have a low vaginal and rectal swab taken which will be processed using the CDC Group B streptococcus guideline. Additionally, a GBS-specific PCR of the swab will be used to identify culture-negative cases of GBS carriage. 5ml of venous blood will be taken from the mother and 5ml of blood taken, after delivery, from the placenta (from the umbilical vein) for GBS antibody studies.

This study will establish the burden of clinical early onset neonatal sepsis in our population. Additionally this study will establish the prevalence of maternal GBS carriage and assess the potential for intrapartum antibiotic prophylaxis for reducing the burden of neonatal sepsis in this setting. It will also define the serotypes and antibiotic susceptibility profile of carried and invasive GBS strains.

ELIGIBILITY:
Part 1. The contribution of GBS to EO neonatal sepsis at Maela Refugee Camp study

1. Infants, < 7 days of age, who are born to mothers who followed antenatal care at SMRU antenatal clinic, Maela Refugee Camp and have a clinical diagnosis of sepsis
2. Written informed consent from the mother

Exclusion criteria:

1. Severe congenital abnormality identified prenatally or at birth
2. Infants less than 28 weeks gestation Part 2. The GBS carriage, seroepidemiology and GBS antibody study

Inclusion criteria:

1. Mothers following antenatal care at SMRU antenatal clinic, Maela camp who are 28 - 30 weeks gestation
2. Written informed consent from the mother

Exclusion criteria:

1. Mothers receiving antibiotics at the time of sampling

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All expectant mothers who follow ANC care at SMRU Maela Refugee Camp and their infants.
Sampling Method: Non-Probability Sample
Enrollment: 849 (Actual)
Dates: Start 2009-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Incidence of early onset neonatal sepsis (including the prevalence of culture positive and culture negative EO GBS sepsis) | 7 days after delivery

SECONDARY OUTCOMES:
Perinatal risk factors for early onset neonatal sepsis | 7 days after delivery
Prevalence of maternal GBS carriage | During labour
GBS serotype specific antibody prevalence | During labour
serotypes and antibiotic susceptibility profile of carried and invasive GBS strains | During labour

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, MD, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

REFERENCES:
- [Result] Turner C, Turner P, Po L, Maner N, De Zoysa A, Afshar B, Efstratiou A, Heath PT, Nosten F. Group B streptococcal carriage, serotype distribution and antibiotic susceptibilities in pregnant women at the time of delivery in a refugee population on the Thai-Myanmar border. BMC Infect Dis. 2012 Feb 8;12:34. doi: 10.1186/1471-2334-12-34. PMID 22316399
- [Result] Turner C, Turner P, Hoogenboom G, Aye Mya Thein N, McGready R, Phakaudom K, De Zoysa A, Efstratiou A, Heath PT, Nosten F. A three year descriptive study of early onset neonatal sepsis in a refugee population on the Thailand Myanmar border. BMC Infect Dis. 2013 Dec 21;13:601. doi: 10.1186/1471-2334-13-601. PMID 24359288